CLINICAL TRIAL: NCT03434379
Title: A Phase III, Open-Label, Randomized Study of Atezolizumab in Combination With Bevacizumab Compared With Sorafenib in Patients With Untreated Locally Advanced or Metastatic Hepatocellular Carcinoma
Brief Title: A Study of Atezolizumab in Combination With Bevacizumab Compared With Sorafenib in Patients With Untreated Locally Advanced or Metastatic Hepatocellular Carcinoma
Acronym: IMbrave150
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YO40245; 2017-003691-31 (EudraCT Number)
Record Dates: First submitted 2018-01-31; First posted 2018-02-15 (Actual); Results first posted 2021-11-05 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab; Sorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atezolizumab + Bevacizumab (Experimental): Participants will receive Atezolizumab + Bevacizumab until unacceptable toxicity or loss of clinical benefit as determined by the investigator
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab
- Sorafenib (Active Comparator): Participants will receive Sorafenib until unacceptable toxicity or loss of clinical benefit as determined by the investigator
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered by IV, 1200 mg on day 1 of each 21 day cycle
  Arms: Atezolizumab + Bevacizumab
Drug: Bevacizumab — Bevacizumab will be administered by IV, 15 mg/kg on day 1 of each 21 day cycle
  Arms: Atezolizumab + Bevacizumab
Drug: Sorafenib — Sorafenib will be administered by mouth, 400 mg twice per day, on days 1-21 of each 21-day cycle
  Arms: Sorafenib

SUMMARY:
This study will evaluate the efficacy and safety of atezolizumab in combination with bevacizumab compared with sorafenib in participants with locally advanced or metastatic Hepatocellular Carcinoma (HCC) who have received no prior systemic treatment.

DETAILED DESCRIPTION:
The participants will be randomized in a 2:1 ratio to one of the two treatment arms: Arm A (experimental arm): Atezolizumab +bevacizumab; Arm B (control arm): Sorafenib

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic and/or unresectable Hepatocellular Carcinoma (HCC)
* No prior systemic therapy for HCC. Previous use of herbal therapies/traditional Chinese medicines with anti-cancer activity included in the label is allowed, provided that these medications are discontinued prior to randomization.
* At least one measurable untreated lesion
* ECOG Performance Status of 0 or 1
* Adequate hematologic and end-organ function
* For women of childbearing potential: agreement to remain abstinent
* For men: agreement to remain abstinent
* Child-Pugh class A

Exclusion Criteria:

* History of leptomeningeal disease
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan
* Known active tuberculosis
* History of malignancy other than HCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within at least 5 months after the last dose of atezolizumab, 6 months after the last dose of bevacizumab, or 1 month after the last dose of sorafenib
* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
* Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high-risk for bleeding
* A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment.
* Moderate or severe ascites
* History of hepatic encephalopathy
* Co-infection of HBV and HCV
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled or symptomatic hypercalcemia
* Treatment with systemic immunostimulatory agents
* Inadequately controlled arterial hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Evidence of bleeding diathesis or significant coagulopathy
* History of intestinal obstruction and/or clinical signs or symptoms of GI obstruction including sub-occlusive disease related to the underlying disease or requirement for routine parenteral hydration
* Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture
* Metastatic disease that involves major airways or blood vessels, or centrally located mediastinal tumor masses
* Local therapy to liver within 28 days prior to initiation of study treatment or non-recovery from side effects of any such procedure
* Chronic daily treatment with a non-steroidal anti-inflammatory drug (NSAID)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (119):
- United States (21):
  - St. Josephs Hospital and Medical Center, Phoenix, Arizona
  - City of Hope, Duarte, California
  - Uni of California - San Diego; Cancer Center & Dept of Medicine, La Jolla, California
  - Kaiser Permanente Northern California, Novato, California
  - University of California Irvine Medical Center, Orange, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - Kaiser Permanente - San Francisco Medical Center, San Francisco, California
  - University of California Los Angeles, Santa Monica, California
  - Kaiser Permanente - Walnut Creek, Walnut Creek, California
  - Banner MD Anderson Cancer Center, Greeley, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Washington University; Wash Uni. Sch. Of Med, St Louis, Missouri
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Laura and ISAAC Perlmutter Cancer Center at NYU Langone., New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - M.D Anderson Cancer Center; Uni of Texas At Houston, Houston, Texas
  - Swedish Cancer Inst., Seattle, Washington
- Australia (4):
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Sunshine Hospital, St Albans, Victoria
- Canada (4):
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Centre hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre - Glen Site, Montreal, Quebec
- China (21):
  - Peking Union Medical College Hospital, Beijing
  - Beijing Friendship Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - the First Hospital of Jilin University, Changchun
  - Jilin Cancer Hospital, Changchun
  - Hunan Cancer Hospital, Changsha
  - The First People's Hospital of Foshan; Local Ethic Committee, Foshan
  - The 900th Hospital of PLA joint service support force, Fuzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou
  - Sir Run Run Shaw Hospital, Hangzhou
  - Zhejiang Cancer Hospital; Zhejiang Cancer Hospital cancer department, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Anhui Province Cancer Hospital, Hefei
  - General Hospital of Jinan Military Command of PLA, Jinan
  - The 81st Hospital of P.L.A., Nanjing
  - Zhongshan Hospital Fudan University, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tongji Hosp, Tongji Med. Col, Huazhong Univ. of Sci. & Tech, Wuhan
- Czechia (2):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
- France (10):
  - Hopital Claude Huriez;Gastro Enterologie, Lille
  - Hopital De La Croix Rousse; Hepatologie Gastro Enterologie, Lyon
  - Hopital Timone Adultes; Gastro Enterologie, Marseille
  - Hopital Saint-Eloi; Hepatologie-Gastro-Enterologie, Montpellier
  - Hopital Hotel Dieu Et Hme; Hepatologie Gastro Enterologie, Nantes
  - CHU Nice - Hôpital de l'Archet 2; service Hepato gastro enterologie, Nice
  - Hopital Charles Nicolle; Gastroenterologie, Rouen
  - Hopital Hautepierre; Gastro Enterologie, Strasbourg
  - Hôpital d'Adultes; Service hépato-gastro-entérologie, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy; Gastro-Enterologie, Villejuif
- Germany (7):
  - Campus Virchow-Klinikum Charité Centrum 13; Medizinische Klinik; Abt.Hepatologie u.Gastroenterologie, Berlin
  - Klinik Johann Wolfgang von Goethe Uni; Zentrum der Inneren Medizin; Medizinische Klinik I, Frankfurt
  - Universitaetsklinikum Hamburg-Eppendorf; I. Medizinische Klinik - Gastroenterologie, Hamburg
  - Med. Hochschule Hannover; Gastroenterologie, Hanover
  - Universitätsklinikum Leipzig Medizinische Klinik II Gastroenterolog. u. Hepatolog., Leipzig
  - Uniklinik Mainz; I. Medizinische Klinik, Mainz
  - Klinikum der Uni Regensburg; Klinik f.Innere Medizin I Abt. Hämatologie und Internistische Onkologie, Regensburg
- Hong Kong (2):
  - Queen Mary Hospital; Dept. Of Haematology & Oncology, Hong Kong
  - Prince of Wales Hosp; Dept. Of Clinical Onc, Shatin
- Italy (6):
  - Az. Osp. Rummo; Oncologia Medica, Benevento, Campania
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - Az. Osp. S. Luigi Gonzaga; Divisione Di Oncologia Medica, Orbassano, Piedmont
  - A.O.U. Cagliari-P.O. Monserrato;U.O. Oncologia, Cagliari, Sardinia
  - Azienda Ospedaliero - Universitaria Pisana U.O. Oncologia Medica 2 Universitaria ? Polo Oncologico, Pisa, Tuscany
  - IRCCS Istituto Oncologico Veneto (IOV); Oncologia Medica Prima, Padua, Veneto
- Japan (13):
  - Chiba University Hospital, Chiba
  - National Cancer Center Hospital East, Chiba
  - Kurume University Hospital, Fukuoka
  - Sapporo Kosei Genaral Hospital, Hokkaido
  - Hokkaido University Hospital, Hokkaido
  - Kanazawa University Hospital, Ishikawa
  - Kitasato University Hospital, Kanagawa
  - Kumamoto University Hospital, Kumamoto
  - Osaka Metropolitan University Hospital, Osaka
  - Kindai University Hospital, Osaka
  - Saga-ken Medical Centre Koseikan, Saga
  - Shizuoka Cancer Center, Shizuoka
  - Japanese Red Cross Musashino Hospital, Tokyo
- Poland (5):
  - Copernicus Podmiot Medyczny Sp. z o.o. Wojewodzkie Centrum Onkologii, Gdansk
  - ID Clinic, Mysłowice
  - SP ZOZ MSWiA z WARMINSKO-MAZURSKIM CENTRUM ONKOLOGII; CLINICAL ONCOLOGY, CLINICAL IMMUNOLOGY, Olsztyn
  - Narodowy Instytut Onkologii im. Marii Sk?odowskiej-Curie - Pa?stwowy Instytut Badawczy, Warsaw
  - Dolno?l?skie Centrum Onkologii; Oddzia? Onkologii Klinicznej i Chemioterapii, Wroc?aw
- Russia (2):
  - FSBI "National Medical Research Center of Oncology N.N. Blokhin?; Clinical Biotechnologies, Moscow, Moscow Oblast
  - GBUZ Saint Petersburg Clinical Research Center of Specialized Types of Care (Oncology), Saint Petersburg, Sankt-Peterburg
- Singapore (2):
  - National Cancer Centre, Singapore
  - Tan Tock Seng Hospital; Oncology, Singapore
- South Korea (6):
  - Chonnam National University Hwasun Hospital, Jeollanam-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan University Hosiptal, Ulsan
- Spain (5):
  - Hospital Universitari Vall d'Hebron; Oncology, Barcelona
  - Hospital Clinico San Carlos; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
  - Centro Integral Oncologico Clara Campal; Servicio de Oncología, Madrid
  - Hospital Universitario Miguel Servet; Servicio de Oncologia Medica, Zaragoza
- Taiwan (5):
  - National Cheng Kung University Hospital; Oncology, Tainan
  - Chi-Mei Medical Centre; Hematology & Oncology, Tainan
  - Veterans General Hospital; Cancer Center, Taipei
  - National Taiwan Uni Hospital; Dept of Oncology, Taipei
  - Chang Gung Memorial Hospital-Linkou; Dept of Oncology, Taoyuan
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Free Hospital; Dept of Oncology, London
  - King'S College Hospital, London
  - Christie Hospital Nhs Trust; Medical Oncology, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Xu XQ, Li WM, Shi LC, Wang H, Li S, Huang C, You H, Jia JD, He YW, Kong YY. Impact of temporary atezolizumab and bevacizumab interruption on survival in advanced HCC: an IMbrave150 analysis. Oncologist. 2025 Sep 1;30(9):oyaf269. doi: 10.1093/oncolo/oyaf269. PMID 40891895
- [Derived] Kaseb AO, Guan Y, Gok Yavuz B, Abbas AR, Lu S, Hasanov E, Toh HC, Verret W, Wang Y. Serum IGF-1 Scores and Clinical Outcomes in the Phase III IMbrave150 Study of Atezolizumab Plus Bevacizumab versus Sorafenib in Patients with Unresectable Hepatocellular Carcinoma. J Hepatocell Carcinoma. 2022 Oct 11;9:1065-1079. doi: 10.2147/JHC.S369951. eCollection 2022. PMID 36254201
- [Derived] Li Y, Liang X, Li H, Chen X. Atezolizumab plus bevacizumab versus nivolumab as first-line treatment for advanced or unresectable hepatocellular carcinoma: A cost-effectiveness analysis. Cancer. 2022 Nov 15;128(22):3995-4003. doi: 10.1002/cncr.34457. Epub 2022 Sep 16. PMID 36111952
- [Derived] Cheng AL, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Lim HY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Ma N, Nicholas A, Wang Y, Li L, Zhu AX, Finn RS. Updated efficacy and safety data from IMbrave150: Atezolizumab plus bevacizumab vs. sorafenib for unresectable hepatocellular carcinoma. J Hepatol. 2022 Apr;76(4):862-873. doi: 10.1016/j.jhep.2021.11.030. Epub 2021 Dec 11. PMID 34902530
- [Derived] Salem R, Li D, Sommer N, Hernandez S, Verret W, Ding B, Lencioni R. Characterization of response to atezolizumab + bevacizumab versus sorafenib for hepatocellular carcinoma: Results from the IMbrave150 trial. Cancer Med. 2021 Aug;10(16):5437-5447. doi: 10.1002/cam4.4090. Epub 2021 Jun 29. PMID 34189869
- [Derived] Galle PR, Finn RS, Qin S, Ikeda M, Zhu AX, Kim TY, Kudo M, Breder V, Merle P, Kaseb A, Li D, Mulla S, Verret W, Xu DZ, Hernandez S, Ding B, Liu J, Huang C, Lim HY, Cheng AL, Ducreux M. Patient-reported outcomes with atezolizumab plus bevacizumab versus sorafenib in patients with unresectable hepatocellular carcinoma (IMbrave150): an open-label, randomised, phase 3 trial. Lancet Oncol. 2021 Jul;22(7):991-1001. doi: 10.1016/S1470-2045(21)00151-0. Epub 2021 May 27. PMID 34051880
- [Derived] Wen F, Zheng H, Zhang P, Liao W, Zhou K, Li Q. Atezolizumab and bevacizumab combination compared with sorafenib as the first-line systemic treatment for patients with unresectable hepatocellular carcinoma: A cost-effectiveness analysis in China and the United states. Liver Int. 2021 May;41(5):1097-1104. doi: 10.1111/liv.14795. Epub 2021 Feb 8. PMID 33556230
- [Derived] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 117 sites in 17 countries: Australia, Canada, China, Czech Republic, Germany, Spain, France, United Kingdom, Hong Kong, Italy, Japan, Republic of Korea, Poland, Russian Federation, Singapore, Taiwan, United States.
Pre-assignment Details: The total study population included 558 participants. The Global population included 501 participants. An additional 57 participants enrolled during the China Extension. The total China population included 137 Chinese participants from the Global population plus 57 participants from the China extension. 137 participants were part of the Global as well as China populations. Separate analyses were performed for the Global population and the China population in the study.
Groups:
- Sorafenib - Global: Participants in the Global population received sorafenib until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
- Atezolizumab + Bevacizumab - Global: Participants in the Global population received Atezolizumab + Bevacizumab until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
- Sorafenib - China: Participants in the China population received sorafenib until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
- Atezolizumab + Bevacizumab - China: Participants in the China population received Atezolizumab + Bevacizumab until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
Period: Global Period
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global | Sorafenib - China | Atezolizumab + Bevacizumab - China
Started | 165 | 336 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 165 | 336 | 0 | 0
Not completed — Lost to Follow-up | 3 | 6 | 0 | 0
Not completed — Death | 115 | 228 | 0 | 0
Not completed — Withdrawal by Subject | 20 | 21 | 0 | 0
Not completed — Reason Unspecified | 0 | 1 | 0 | 0
Not completed — Study Ended by Sponsor | 26 | 80 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Period: China Extension Period
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global | Sorafenib - China | Atezolizumab + Bevacizumab - China
Started | 0 | 0 | 61 (n=43 Chinese participants from the sorafenib Global population are included in the China population.) | 133 (n=94 Chinese participants from the Atezolizumab + Bevacizumab Global population are included in the China population.)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 61 | 133
Not completed — Lost to Follow-up | 0 | 0 | 2 | 3
Not completed — Death | 0 | 0 | 46 | 88
Not completed — Withdrawal by Subject | 0 | 0 | 8 | 6
Not completed — Study Ended by Sponsor | 0 | 0 | 5 | 36

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included 558 participants (All) with 501 in the Global population. An additional 57 participants enrolled in the China Extension. The China population included 137 Chinese participants from the Global population plus 57 participants from the China Extension. The Global population and China population were analyzed separately.
Groups:
- Sorafenib - All: All participants either in the Global or China population received sorafenib until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
- Atezolizumab + Bevacizumab - All: All participants either in the Global or China population received Atezolizumab + Bevacizumab until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
- Total: Total of all reporting groups
Arm/Group | Sorafenib - All | Atezolizumab + Bevacizumab - All | Total
Number analyzed (Participants) | 183 | 375 | 558
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The Global population included 501 participants. The China population included 57 participants enrolled during the China Extension plus 137 Chinese participants from the Global population.
  years
    Global: number analyzed (Participants) | 165 | 336 | 501
    Global | 64.4 (10.9) | 62.9 (11.9) | 63.4 (11.6)
    China: number analyzed (Participants) | 61 | 133 | 194
    China | 57.5 (12.7) | 55.3 (12.0) | 56.0 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Global population included 501 participants. The China population included 57 participants enrolled during the China Extension plus 137 Chinese participants from the Global population.
  Participants
    Global: number analyzed (Participants) | 165 | 336 | 501
    Global: Female | 28 | 59 | 87
    Global: Male | 137 | 277 | 414
    China: number analyzed (Participants) | 61 | 133 | 194
    China: Female | 12 | 17 | 29
    China: Male | 49 | 116 | 165
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Global population included 501 participants. The China population included 57 participants enrolled during the China Extension plus 137 Chinese participants from the Global population.
  Participants
    Global: number analyzed (Participants) | 165 | 336 | 501
    Global: Hispanic or Latino | 4 | 9 | 13
    Global: Not Hispanic or Latino | 149 | 306 | 455
    Global: Unknown or Not Reported | 12 | 21 | 33
    China: number analyzed (Participants) | 61 | 133 | 194
    China: Hispanic or Latino | 0 | 0 | 0
    China: Not Hispanic or Latino | 61 | 133 | 194
    China: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Global population included 501 participants. The China population included 57 participants enrolled during the China Extension plus 137 Chinese participants from the Global population.
  Participants
    Global: number analyzed (Participants) | 165 | 336 | 501
    Global: American Indian or Alaska Native | 1 | 0 | 1
    Global: Asian | 96 | 188 | 284
    Global: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Global: Black or African American | 4 | 6 | 10
    Global: White | 52 | 123 | 175
    Global: More than one race | 0 | 0 | 0
    Global: Unknown or Not Reported | 12 | 19 | 31
    China: number analyzed (Participants) | 61 | 133 | 194
    China: American Indian or Alaska Native | 0 | 0 | 0
    China: Asian | 61 | 133 | 194
    China: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    China: Black or African American | 0 | 0 | 0
    China: White | 0 | 0 | 0
    China: More than one race | 0 | 0 | 0
    China: Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in the Global Population
Description: OS was defined as the time from randomization to death from any cause.
Time Frame: From randomization to death from any cause up to the clinical cut off date (CCOD) of 29Aug2019 (up to approximately 18 months) and 31Aug2020 (up to approximately 30 months)
Population: Global ITT population consisted of all randomized participants in the Global population, whether or not the participant had received the assigned study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 165 | 336
months
  At CCOD 18 months | 13.24 [10.41 to NA] — NA = not estimable due to the limited number of events observed | NA [NA to NA] — NA = not estimable due to the limited number of events observed
  At CCOD 30 months | 13.40 [11.37 to 16.85] | 19.22 [17.02 to 23.66]
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; At CCOD 18 months; Stratified by geographic region (Asia [excluding Japan] vs. rest of world), macrovascular invasion and/or extrahepatic spread (presence vs. absence), and baseline alpha-fetoprotein (AFP: <400 vs. >/= 400 ng/mL); Test type: Superiority; p = 0.0006, Log Rank; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.42 to 0.79]
Statistical Analysis 2: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; At CCOD 30 months; Stratified by geographic region (Asia [excluding Japan] vs. rest of world), macrovascular invasion and/or extrahepatic spread (presence vs. absence), and baseline alpha-fetoprotein (AFP: <400 vs. >/= 400 ng/mL); Test type: Superiority; p = 0.0009, Log Rank; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.52 to 0.85]

2. Primary Outcome: Progression Free Survival by Independent Review Facility-Assessment (PFS-IRF) Per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 in the Global Population
Description: PFS was defined as the time from randomization to the first occurrence of progressive disease (PD) or death from any cause whichever occurs first as determined by an IRF according to RECIST v1.1. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 millimeters (mm).
Time Frame: Randomization to the first occurrence of disease progression or death from any cause up to CCOD of 29Aug2019 (up to approximately 18 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 165 | 336
months | 4.27 [3.98 to 5.55] | 6.83 [5.75 to 8.28]
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; Stratified by geographic region (Asia [excluding Japan] vs. rest of world), macrovascular invasion and/or extrahepatic spread (presence vs. absence), and baseline AFP (<400 vs. >/= 400 ng/mL); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.47 to 0.76]

3. Primary Outcome: Overall Survival (OS) in the China Population
Description: OS was defined as the time from randomization to death from any cause.
Time Frame: as for outcome 1
Population: China ITT population consisted of all randomized participants in the China population, whether or not the participant had received the assigned study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - China | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 61 | 133
months
  At CCOD 18 months | 11.37 [6.74 to NA] — NA = not estimable due to the limited number of events observed | NA [13.50 to NA] — NA = not estimable due to the limited number of events observed
  At CCOD 30 months | 11.37 [6.74 to 16.07] | 24.05 [17.12 to NA] — NA = not estimable due to the limited number of events observed
Statistical Analysis 1: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; At CCOD 18 months; Stratified by macrovascular invasion and/or extrahepatic spread (presence vs. absence), and baseline AFP (<400 vs. >/= 400 ng/mL); Test type: Superiority; p = 0.0026, Log Rank; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.25 to 0.76]
Statistical Analysis 2: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; At CCOD 30 months; Stratified by macrovascular invasion and/or extrahepatic spread (presence vs. absence), and baseline AFP (<400 vs. >/= 400 ng/mL); Test type: Superiority; p = 0.0019, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.35 to 0.80]

4. Primary Outcome: PFS-IRF Per RECIST v1.1 in the China Population
Description: as for outcome 2
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - China | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 61 | 133
months | 3.19 [2.56 to 4.76] | 5.72 [4.17 to 8.28]
Statistical Analysis 1: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; Stratified by macrovascular invasion and/or extrahepatic spread (presence vs. absence), and baseline AFP (<400 vs. >/= 400 ng/mL); Test type: Superiority; p = 0.0117, Log Rank; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.40 to 0.90]

5. Secondary Outcome: Objective Response Rate by IRF-Assessment (ORR-IRF) Per RECIST v1.1 in the Global Population
Description: ORR was defined as the percentage of participants with a complete response (CR) or a partial response (PR) as determined by the IRF according to RECIST v1.1. CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. OR=CR+PR
Time Frame: Randomization up to CCOD of 29Aug2019 (up to approximately 18 months)
Population: Global ITT population with measurable disease at baseline consisted of all randomized participants in the Global population, whether or not the participant had received the assigned study treatment, and had measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 159 | 326
percentage of participants | 11.9 [7.35 to 18.03] | 27.3 [22.54 to 32.48]
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.90, 95% CI 2-sided [1.68 to 5.01]

6. Secondary Outcome: Objective Response Rate by IRF-Assessment (ORR-IRF) Per Hepatocellular Carcinoma (HCC) Modified RECIST (mRECIST) in the Global Population
Description: ORR was defined as the percentage of participants with CR or PR as determined by the IRF according to HCC mRECIST. HCC mRECIST differentiates between vital tumor and necrotic areas in the liver measuring only the residual vital tumor mass in the liver. CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. OR=CR+PR
Time Frame: Randomization up to CCOD of 29Aug2019 (up to approximately 18 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 158 | 325
percentage of participants | 13.3 [8.42 to 19.60] | 33.2 [28.13 to 38.64]
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.39, 95% CI 2-sided [2.02 to 5.71]

7. Secondary Outcome: ORR by Investigator-Assessment (ORR-INV) Per RECIST v1.1 in the Global Population
Description: ORR was defined as the percentage of participants with CR or PR as determined by the investigator according to RECIST v1.1. CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. OR=CR+PR
Time Frame: Randomization up to CCOD of 29Aug2019 (up to approximately 18 months)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 164 | 336
percentage of participants | 5.5 [2.54 to 10.16] | 25.6 [21.01 to 30.61]
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 6.15, 95% CI 2-sided [2.99 to 12.66]

8. Secondary Outcome: Duration of Response by IRF-Assessment (DOR-IRF) Per RECIST v1.1 in the Global Population
Description: DOR was defined as the time interval from the date of first occurrence of a documented objective response (CR or PR, whichever status is recorded first) until the first date that disease progression (PD) or death was documented, whichever occurs first as determined by the IRF according to RECIST v1.1. CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 mm.
Time Frame: Randomization up to CCOD of 29Aug2019 (up to approximately 18 months)
Population: The analysis population included Global participants with a confirmed response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 19 | 89
months | 6.28 [4.67 to NA] — NA = not estimable due to the limited number of events observed | NA [NA to NA] — NA = not estimable due to the limited number of events observed
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0051, Log Rank; Hazard Ratio (HR) = 0.23, 95% CI 2-sided [0.08 to 0.70]

9. Secondary Outcome: Duration of Response by IRF Assessment (DOR-IRF) Per HCC mRECIST in the Global Population
Description: DOR was defined as the time interval from the date of first occurrence of a documented objective response (CR or PR, whichever status is recorded first) until the first date that disease progression (PD) or death was documented, whichever occurs first as determined by the IRF according to HCC mRECIST. HCC mRECIST differentiates between vital tumor and necrotic areas in the liver, measuring only the residual vital tumor mass in the liver CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 mm.
Time Frame: Randomization up to CCOD of 29Aug2019 (up to approximately 18 months)
Population: The analysis population included Global participants with a confirmed response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 21 | 108
months | 6.28 [4.86 to NA] — NA = not estimable due to the limited number of events observed | NA [NA to NA] — NA = not estimable due to the limited number of events observed
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0048, Log Rank; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.12 to 0.73]

10. Secondary Outcome: Duration of Response by Investigator Assessment (DOR-INV) Per RECIST v1.1 in the Global Population
Description: DOR was defined as the time interval from the date of first occurrence of a documented objective response (CR or PR, whichever status is recorded first) until the first date that disease progression (PD) or death was documented, whichever occurs first as determined by the investigator according to RECIST v1.1. CR: disappearance of all target lesions. PR: At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 mm.
Time Frame: Randomization up to CCOD of 29Aug2019 (up to approximately 18 months)
Population: The analysis population included Global participants with a confirmed response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 9 | 86
months | NA [5.39 to NA] — NA = not estimable due to the limited number of events observed | 13.08 [13.08 to NA] — NA = not estimable due to the limited number of events observed
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.4187, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.16 to 2.15]

11. Secondary Outcome: PFS-IRF Per HCC mRECIST in the Global Population
Description: PFS was defined as the time from randomization to the first occurrence of progressive disease or death from any cause whichever occurs first as determined by the IRF according to HCC mRECIST. HCC mRECIST differentiates between vital tumor and necrotic areas in the liver, measuring only the residual vital tumor mass in the liver. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 millimeters (mm).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 165 | 336
months | 4.24 [3.98 to 5.45] | 6.83 [5.72 to 7.69]
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.46 to 0.74]

12. Secondary Outcome: PFS by Investigator Assessment (PFS-INV) Per RECIST v1.1 in the Global Population
Description: PFS was defined as the time from randomization to the first occurrence of progressive disease or death from any cause whichever occurs first as determined by the investigator according to RECIST v1.1. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 millimeters (mm).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 165 | 336
months | 2.89 [2.76 to 4.17] | 7.06 [5.68 to 8.44]
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.36 to 0.57]

13. Secondary Outcome: Time to Progression (TTP) by IRF Assessment (TTP-IRF) Per RECIST v1.1 in the Global Population
Description: Time to progression was defined as the time from the date of randomization to the date of the first documented tumor progression as determined by the IRF according to RECIST v1.1. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 millimeters (mm).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 165 | 336
months | 5.59 [4.21 to 7.72] | 8.57 [6.83 to 9.86]
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0105, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.53 to 0.92]

14. Secondary Outcome: TTP-IRF Per HCC mRECIST in the Global Population
Description: Time to progression was defined as the time from the date of randomization to the date of the first documented tumor progression as determined by the IRF according to HCC mRECIST. HCC mRECIST differentiates between vital tumor and necrotic areas in the liver, measuring only the residual vital tumor mass in the liver. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 millimeters (mm).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 165 | 336
months | 5.55 [4.21 to 7.69] | 8.28 [6.80 to 9.86]
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0063, Log Rank; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.52 to 0.90]

15. Secondary Outcome: TTP by Investigator Assessment (TTP-INV) Per RECIST v1.1 in the Global Population
Description: Time to progression was defined as the time from the date of randomization to the date of the first documented tumor progression as determined by the investigator according to RECIST v1.1. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 millimeters (mm).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 165 | 336
months | 3.98 [2.83 to 4.30] | 8.54 [6.93 to 9.92]
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.35 to 0.57]

16. Secondary Outcome: Overall Survival by Baseline AFP in the Global Population
Description: OS was defined as the time from randomization to death from any cause. Subpopulations with baseline AFP <400 ng/mL and AFP>/= 400 ng/mL were analyzed.
Time Frame: From randomization to death from any cause up to CCOD of 29Aug2019 (up to approximately 18 months)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 165 | 336
months
  AFP <400 ng/mL: number analyzed (Participants) | 104 | 210
  AFP <400 ng/mL | 13.93 [11.73 to NA] — NA = not estimable due to the limited number of events observed | NA [NA to NA] — NA = not estimable due to the limited number of events observed
  AFP >/=400 ng/mL: number analyzed (Participants) | 61 | 126
  AFP >/=400 ng/mL | 9.10 [5.75 to NA] — NA = not estimable due to the limited number of events observed | 12.78 [10.15 to NA] — NA = not estimable due to the limited number of events observed
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; AFP <400 ng/mL and stratified by geographic region (Asia [excluding Japan] vs. rest of world), macrovascular invasion and/or extrahepatic spread (presence vs. absence); Test type: Superiority; p = 0.0019, Log Rank; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.32 to 0.78]
Statistical Analysis 2: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; AFP >/= 400 ng/mL and stratified by geographic region (Asia [excluding Japan] vs. rest of world), macrovascular invasion and/or extrahepatic spread (presence vs. absence); Test type: Superiority; p = 0.0879, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.42 to 1.06]

17. Secondary Outcome: PFS-IRF Per RECIST v1.1 by Baseline AFP in the Global Population
Description: PFS was defined as the time from randomization to the first occurrence of progressive disease or death from any cause whichever occurs first as determined by the IRF according to RECIST v1.1. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 millimeters (mm). Subpopulations with baseline AFP <400 ng/mL and AFP>/= 400 ng/mL were analyzed.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 165 | 336
months
  AFP <400 ng/mL: number analyzed (Participants) | 104 | 210
  AFP <400 ng/mL | 4.40 [4.01 to 6.21] | 8.28 [6.83 to 11.04]
  AFP >/=400 ng/mL: number analyzed (Participants) | 61 | 126
  AFP >/=400 ng/mL | 4.14 [2.76 to 5.26] | 5.19 [3.94 to 6.77]
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; AFP<400 ng/mL and stratified by geographic region (Asia [excluding Japan] vs. rest of world), macrovascular invasion and/or extrahepatic spread (presence vs. absence); Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.37 to 0.68]
Statistical Analysis 2: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; AFP >/=400 ng/mL and stratified by geographic region (Asia [excluding Japan] vs. rest of world), macrovascular invasion and/or extrahepatic spread (presence vs. absence); Test type: Superiority; p = 0.2159, Log Rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.53 to 1.15]

18. Secondary Outcome: PFS-INV Per RECIST v1.1 by Baseline AFP in the Global Population
Description: PFS was defined as the time from randomization to the first occurrence of progressive disease or death from any cause whichever occurs first as determined by the investigator according to RECIST v1.1. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of >/= 5 millimeters (mm). Subpopulations with baseline AFP <400 ng/mL and AFP>/= 400 ng/mL were analyzed.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 165 | 336
months
  AFP <400 ng/mL: number analyzed (Participants) | 104 | 210
  AFP <400 ng/mL | 3.98 [2.79 to 5.62] | 8.41 [7.06 to 9.66]
  AFP >/=400 ng/mL: number analyzed (Participants) | 61 | 126
  AFP >/=400 ng/mL | 2.79 [1.58 to 3.98] | 5.42 [4.17 to 6.90]
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.31 to 0.57]
Statistical Analysis 2: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; [analysis description as in outcome 17, analysis 2]; Test type: Superiority; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.35 to 0.73]

19. Secondary Outcome: Time to Deterioration (TTD) in the Global Population
Description: TTD was defined as the time from randomization to the first deterioration (decrease from baseline of >/= 10 points) in the patient-reported health-related global health status/quality of life (GHS /HRQoL), physical function or role function scales of the European Organization for Research and Treatment of Cancer quality-of-life questionnaire for cancer (EORTC) QLQ-C30, maintained for two consecutive assessments, or one assessment followed by death from any cause within 3 weeks.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 165 | 336
months
  Physical Functioning | 4.86 [3.48 to 6.24] | 13.14 [9.69 to NA] — NA = not estimable due to the limited number of events observed
  Role Functioning | 3.58 [2.20 to 5.98] | 9.13 [6.51 to NA] — NA = not estimable due to the limited number of events observed
  GHS/QoL | 3.58 [3.02 to 6.97] | 11.24 [5.98 to NA] — NA = not estimable due to the limited number of events observed
Statistical Analysis 1: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; Physical Functioning: Stratified by geographic region (Asia [excluding Japan] vs. rest of world), macrovascular invasion and/or extrahepatic spread (presence vs. absence), and baseline AFP (<400 vs. >/= 400 ng/mL); Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.39 to 0.73]
Statistical Analysis 2: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; Role Functioning: Stratified by geographic region (Asia [excluding Japan] vs. rest of world), macrovascular invasion and/or extrahepatic spread (presence vs. absence), and baseline AFP (<400 vs. >/= 400 ng/mL); Test type: Superiority; p = 0.0019, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.46 to 0.84]
Statistical Analysis 3: Comparison: Sorafenib - Global vs Atezolizumab + Bevacizumab - Global; GHS/QoL: Stratified by geographic region (Asia [excluding Japan] vs. rest of world), macrovascular invasion and/or extrahepatic spread (presence vs. absence), and baseline AFP (<400 vs. >/= 400 ng/mL); Test type: Superiority; p = 0.0028, Log Rank; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.46 to 0.85]

20. Secondary Outcome: Number of Participants With Adverse Events (AEs) in the Global Population
Description: An adverse event is any untoward medical occurrence in a subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to end of study (up to approximately 56 months)
Population: Global safety population included all randomized Global participants who received any amount of study drug with participants grouped according to the treatment the participant actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 156 | 329
Participants | 154 | 322

21. Secondary Outcome: Maximum Serum Concentration (Cmax) of Atezolizumab at Cycle 1 in the Global Population
Time Frame: Post-dose on Day 1 of Cycle 1 (cycle length = 21 days)
Population: The Global pharmacokinetic (PK)-evaluable population was defined as all participants in the Global population who received any dose of study treatment and who had at least one post-baseline PK sample available.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (mcg/mL)
Arm/Group | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 309
micrograms/milliliter (mcg/mL) | 398 (132)

22. Secondary Outcome: Trough Serum Concentration (Cmin) of Atezolizumab in the Global Population
Time Frame: Pre-dose on Day 1 of Cycles 2, 3, 4, 8, 12 and 16 (cycle length = 21 days)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 329
mcg/mL
  Pre-dose Cycle 2, Day 1: number analyzed (Participants) | 298
  Pre-dose Cycle 2, Day 1 | 79.2 (50.2)
  Pre-dose Cycle 3, Day 1: number analyzed (Participants) | 41
  Pre-dose Cycle 3, Day 1 | 101 (55.4)
  Pre-dose Cycle 4, Day 1: number analyzed (Participants) | 263
  Pre-dose Cycle 4, Day 1 | 131 (63.7)
  Pre-dose Cycle 8, Day 1: number analyzed (Participants) | 134
  Pre-dose Cycle 8, Day 1 | 145 (61.7)
  Pre-dose Cycle 12, Day 1: number analyzed (Participants) | 153
  Pre-dose Cycle 12, Day 1 | 168 (82.9)
  Pre-dose Cycle 16, Day 1: number analyzed (Participants) | 124
  Pre-dose Cycle 16, Day 1 | 167 (65.0)

23. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADAs) to Atezolizumab in the Global Population
Time Frame: Baseline and post-baseline on Day 1 (pre-dose) of Cycles 2, 3, 4, 8, 12, 16 (cycle length = 21 days) and treatment discontinuation visit (up to approximately 30 months)
Population: The Global ADA-evaluable population was defined as all participants in the Global population who received any dose of atezolizumab and who had at least one post-baseline ADA assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 329
percentage of participants
  Baseline: number analyzed (Participants) | 316
  Baseline | 2.2
  Post-baseline: number analyzed (Participants) | 318
  Post-baseline | 29.6

24. Secondary Outcome: Objective Response Rate by IRF-Assessment (ORR-IRF) Per RECIST v1.1 in the China Population
Description: as for outcome 5
Time Frame: Randomization up to CCOD of 29Aug2019 (up to approximately 18 months)
Population: China ITT population with measurable disease at baseline consisted of all randomized participants in the China population, whether or not the participant had received the assigned study treatment, and had measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib - China | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 60 | 130
percentage of participants | 6.7 [1.85 to 16.20] | 24.6 [17.49 to 32.94]
Statistical Analysis 1: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0036, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.60, 95% CI 2-sided [1.53 to 13.86]

25. Secondary Outcome: Objective Response Rate by IRF-Assessment (ORR-IRF) Per Hepatocellular Carcinoma (HCC) Modified RECIST (mRECIST) in the China Population
Description: as for outcome 6
Time Frame: Randomization up to CCOD of 29Aug2019 (up to approximately 18 months)
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib - China | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 59 | 128
percentage of participants | 8.5 [2.81 to 18.68] | 29.7 [21.94 to 38.40]
Statistical Analysis 1: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0013, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.71, 95% CI 2-sided [1.72 to 12.87]

26. Secondary Outcome: ORR by Investigator-Assessment (ORR-INV) Per RECIST v1.1 in the China Population
Description: as for outcome 7
Time Frame: Randomization up to CCOD of 29Aug2019 (up to approximately 18 months)
Population: as for outcome 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sorafenib - China | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 61 | 133
percentage of participants | 4.9 [1.03 to 13.71] | 21.1 [14.47 to 28.97]
Statistical Analysis 1: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0052, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.05, 95% CI 2-sided [1.47 to 17.39]

27. Secondary Outcome: Duration of Response by IRF-Assessment (DOR-IRF) Per RECIST v1.1 in the China Population
Description: as for outcome 8
Time Frame: Randomization up to CCOD of 29Aug2019 (up to approximately 18 months)
Population: The analysis population included China participants with a confirmed response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - China | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 4 | 32
months | NA [4.86 to NA] — NA = not estimable due to the limited number of events observed | NA [8.15 to NA] — NA = not estimable due to the limited number of events observed
Statistical Analysis 1: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.4581, Log Rank; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.02 to 5.85]

28. Secondary Outcome: Duration of Response by IRF Assessment (DOR-IRF) Per HCC mRECIST in the China Population
Description: as for outcome 9
Time Frame: Randomization up to CCOD of 29Aug2019 (up to approximately 18 months)
Population: The analysis population included China participants with a confirmed response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - China | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 5 | 38
months | 4.86 [4.47 to NA] — NA = not estimable due to the limited number of events observed | NA [8.15 to NA] — NA = not estimable due to the limited number of events observed
Statistical Analysis 1: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0100, Log Rank; Hazard Ratio (HR) = 0.08, 95% CI 2-sided [0.01 to 0.91] — Lower limit: <0.01

29. Secondary Outcome: Duration of Response by Investigator Assessment (DOR-INV) Per RECIST v1.1 in the China Population
Description: as for outcome 10
Time Frame: Randomization up to CCOD of 29Aug2019 (up to approximately 18 months)
Population: The analysis population included China participants with a confirmed response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - China | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 3 | 28
months | 5.55 [4.17 to NA] — NA = not estimable due to the limited number of events observed | NA [NA to NA] — NA = not estimable due to the limited number of events observed
Statistical Analysis 1: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.3477, Log Rank; Hazard Ratio (HR) = 0.33, 95% CI 2-sided [0.03 to 3.69]

30. Secondary Outcome: PFS-IRF Per HCC mRECIST in the China Population
Description: as for outcome 11
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - China | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 61 | 133
months | 3.19 [2.56 to 4.76] | 5.72 [4.17 to 8.11]
Statistical Analysis 1: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0103, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.40 to 0.89]

31. Secondary Outcome: PFS by Investigator Assessment (PFS-INV) Per RECIST v1.1 in the China Population
Description: as for outcome 12
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - China | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 61 | 133
months | 2.83 [2.73 to 3.98] | 5.55 [4.21 to 8.34]
Statistical Analysis 1: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.33 to 0.71]

32. Secondary Outcome: Time to Progression (TTP) by IRF Assessment (TTP-IRF) Per RECIST v1.1 in the China Population
Description: as for outcome 13
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - China | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 61 | 133
months | 4.14 [2.76 to 10.15] | 7.00 [5.45 to 9.49]
Statistical Analysis 1: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0927, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.43 to 1.07]

33. Secondary Outcome: TTP-IRF Per HCC mRECIST in the China Population
Description: as for outcome 14
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - China | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 61 | 133
months | 4.14 [2.76 to 10.15] | 7.00 [5.45 to 9.49]
Statistical Analysis 1: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0861, Log Rank; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.43 to 1.06]

34. Secondary Outcome: TTP by Investigator Assessment (TTP-INV) Per RECIST v1.1 in the China Population
Description: as for outcome 15
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - China | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 61 | 133
months | 2.83 [2.79 to 4.17] | 6.83 [5.32 to 9.33]
Statistical Analysis 1: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.0004, Log Rank; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.33 to 0.74]

35. Secondary Outcome: Time to Deterioration (TTD) in the China Population
Description: as for outcome 19
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib - China | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 61 | 133
months
  Physical Functioning | 5.62 [2.10 to NA] — NA = not estimable due to the limited number of events observed | 13.14 [9.69 to NA] — NA = not estimable due to the limited number of events observed
  Role Functioning | NA [2.14 to NA] — NA = not estimable due to the limited number of events observed | NA [7.20 to NA] — NA = not estimable due to the limited number of events observed
  GHS/QoL | 3.58 [1.48 to 9.82] | 9.76 [6.24 to NA] — NA = not estimable due to the limited number of events observed
Statistical Analysis 1: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; Physical Functioning: Stratified by macrovascular invasion and/or extrahepatic spread (presence vs. absence), and baseline AFP (<400 vs. >/= 400 ng/mL); Test type: Superiority; p = 0.0035, Log Rank; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.26 to 0.78]
Statistical Analysis 2: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; Role Functioning: Stratified by macrovascular invasion and/or extrahepatic spread (presence vs. absence), and baseline AFP (<400 vs. >/= 400 ng/mL); Test type: Superiority; p = 0.2214, Log Rank; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.42 to 1.23]
Statistical Analysis 3: Comparison: Sorafenib - China vs Atezolizumab + Bevacizumab - China; GHS/QoL: Stratified by macrovascular invasion and/or extrahepatic spread (presence vs. absence), and baseline AFP (<400 vs. >/= 400 ng/mL); Test type: Superiority; p = 0.0135, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.32 to 0.88]

36. Secondary Outcome: Number of Participants With Adverse Events (AEs) in the China Population
Description: as for outcome 20
Time Frame: Up to end of study (up to approximately 56 months)
Population: China safety population included all randomized China participants who received any amount of study drug with participants grouped according to the treatment the participant actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib - China | Atezolizumab + Bevacizumab - Global
Number analyzed (Participants) | 58 | 132
Participants | 56 | 131

37. Secondary Outcome: Maximum Serum Concentration (Cmax) of Atezolizumab in the China Population
Time Frame: Post-dose on Day 1 of Cycle 1 (cycle length = 21 days)
Population: The China PK-evaluable population was defined as all participants in the China population who received any dose of study treatment and who had at least one post-baseline PK sample available.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 85
mcg/mL | 456 (153)

38. Secondary Outcome: Trough Serum Concentration (Cmin) of Atezolizumab in the China Population
Time Frame: Pre-dose on Day 1 of Cycles 2, 3, 4, 8, 12 and 16 (cycle length = 21 days)
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 132
mcg/mL
  Pre-dose Cycle 2, Day 1: number analyzed (Participants) | 87
  Pre-dose Cycle 2, Day 1 | 92.6 (65.7)
  Pre-dose Cycle 3, Day 1: number analyzed (Participants) | 4
  Pre-dose Cycle 3, Day 1 | 105 (36.8)
  Pre-dose Cycle 4, Day 1: number analyzed (Participants) | 80
  Pre-dose Cycle 4, Day 1 | 143 (61.4)
  Pre-dose Cycle 8, Day 1: number analyzed (Participants) | 11
  Pre-dose Cycle 8, Day 1 | 177 (61.9)
  Pre-dose Cycle 12, Day 1: number analyzed (Participants) | 20
  Pre-dose Cycle 12, Day 1 | 201 (97.6)
  Pre-dose Cycle 16, Day 1: number analyzed (Participants) | 13
  Pre-dose Cycle 16, Day 1 | 208 (79.4)

39. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADAs) to Atezolizumab in the China Population
Time Frame: Baseline and post-baseline on Day 1 (pre-dose) of Cycles 2, 3, 4, 8, 12, 16 (cycle length = 21 days) and treatment discontinuation visit (up to approximately 18 months)
Population: The China ADA-evaluable population was defined as all participants in the China population who received any dose of atezolizumab and who had at least one post-baseline ADA assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Atezolizumab + Bevacizumab - China
Number analyzed (Participants) | 132
percentage of participants
  Baseline: number analyzed (Participants) | 90
  Baseline | 1.1
  Post-baseline: number analyzed (Participants) | 89
  Post-baseline | 20.2

ADVERSE EVENTS:
Time Frame: Up to end of study (up to approximately 56 months)
Description: All-cause mortality is reported for deaths that occurred during the study based on the ITT population, which included all randomized participants. Serious and other adverse events were reported based on the safety population, which included all randomized participants who received any amount of study drug with participants grouped according to the treatment the participant actually received. Global and China extension periods were analyzed separately.
Arm/Group | Sorafenib - Global | Atezolizumab + Bevacizumab - Global | Sorafenib - China | Atezolizumab + Bevacizumab - China
All-Cause Mortality (participants affected / at risk) | 115/165 | 228/336 | 46/61 | 88/133
Serious Adverse Events (participants affected / at risk) | 51/156 | 171/329 | 12/58 | 54/132
Other Adverse Events (participants affected / at risk) | 147/156 | 311/329 | 55/58 | 129/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib - Global (N=156) | Atezolizumab + Bevacizumab - Global (N=329) | Sorafenib - China (N=58) | Atezolizumab + Bevacizumab - China (N=132)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 5 (7) | 1 (1) | 3 (3)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 2 (4) | 2 (2) | 1 (3)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0) | 2 (2)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Addison's disease (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 2 (2) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 13 (18) | 0 (0) | 6 (9)
Colitis (Gastrointestinal disorders) | 1 (1) | 5 (5) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gastric mucosal lesion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (4) | 11 (11) | 0 (0) | 3 (3)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 10 (12) | 0 (0) | 2 (3)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (5) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 5 (5) | 1 (1) | 5 (5)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 11 (15) | 1 (1) | 4 (7)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 4 (6) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 5 (5)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatorenal failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burkholderia pseudomallei infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis E (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritoneal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 5 (5) | 0 (0) | 3 (3)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 8 (9) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 4 (6) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 7 (7) | 1 (1) | 2 (2)
General physical condition abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Granulocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 3 (3) | 5 (6) | 0 (0) | 1 (2)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural hygroma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VIth nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 3 (4) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal haematoma (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5) | 0 (0) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersplenism (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Scrotal dermatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib - Global (N=156) | Atezolizumab + Bevacizumab - Global (N=329) | Sorafenib - China (N=58) | Atezolizumab + Bevacizumab - China (N=132)
Anaemia (Blood and lymphatic system disorders) | 14 (15) | 38 (56) | 8 (9) | 26 (44)
Leukopenia (Blood and lymphatic system disorders) | 4 (6) | 21 (33) | 4 (6) | 19 (32)
Neutropenia (Blood and lymphatic system disorders) | 4 (7) | 20 (28) | 3 (6) | 12 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (9) | 32 (45) | 5 (5) | 22 (41)
Hypothyroidism (Endocrine disorders) | 3 (3) | 35 (41) | 1 (1) | 15 (19)
Abdominal distension (Gastrointestinal disorders) | 5 (5) | 26 (27) | 4 (4) | 16 (17)
Abdominal pain (Gastrointestinal disorders) | 27 (31) | 50 (63) | 10 (15) | 19 (24)
Abdominal pain upper (Gastrointestinal disorders) | 9 (10) | 20 (30) | 4 (4) | 7 (8)
Ascites (Gastrointestinal disorders) | 8 (10) | 31 (36) | 2 (3) | 9 (10)
Constipation (Gastrointestinal disorders) | 25 (27) | 58 (63) | 5 (5) | 18 (20)
Diarrhoea (Gastrointestinal disorders) | 79 (107) | 75 (109) | 26 (38) | 20 (28)
Nausea (Gastrointestinal disorders) | 25 (28) | 49 (64) | 7 (9) | 18 (22)
Stomatitis (Gastrointestinal disorders) | 7 (7) | 19 (21) | 2 (2) | 4 (4)
Vomiting (Gastrointestinal disorders) | 14 (14) | 34 (49) | 5 (5) | 15 (25)
Asthenia (General disorders) | 21 (23) | 28 (40) | 3 (3) | 11 (12)
Fatigue (General disorders) | 30 (32) | 76 (92) | 6 (6) | 17 (22)
Oedema peripheral (General disorders) | 6 (6) | 45 (55) | 3 (3) | 13 (18)
Pyrexia (General disorders) | 15 (22) | 58 (83) | 6 (9) | 23 (32)
Nasopharyngitis (Infections and infestations) | 4 (4) | 20 (26) | 1 (1) | 7 (10)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 24 (27) | 2 (2) | 22 (26)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 33 (40) | 0 (0) | 13 (13)
Alanine aminotransferase increased (Investigations) | 14 (18) | 56 (80) | 12 (18) | 30 (52)
Aspartate aminotransferase increased (Investigations) | 28 (32) | 77 (116) | 19 (23) | 41 (76)
Blood alkaline phosphatase increased (Investigations) | 11 (12) | 33 (43) | 7 (9) | 19 (29)
Blood bilirubin increased (Investigations) | 23 (27) | 59 (114) | 14 (16) | 35 (86)
Blood creatinine increased (Investigations) | 1 (1) | 20 (32) | 0 (0) | 10 (18)
Platelet count decreased (Investigations) | 18 (22) | 48 (87) | 10 (11) | 27 (65)
Weight decreased (Investigations) | 15 (18) | 50 (55) | 6 (9) | 21 (23)
White blood cell count decreased (Investigations) | 9 (24) | 21 (76) | 9 (15) | 23 (83)
Decreased appetite (Metabolism and nutrition disorders) | 39 (50) | 68 (78) | 12 (15) | 27 (32)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (5) | 23 (40) | 0 (0) | 13 (30)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 (13) | 42 (53) | 5 (8) | 32 (44)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (13) | 13 (19) | 11 (13) | 13 (22)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (7) | 26 (32) | 4 (4) | 9 (16)
Hypophosphataemia (Metabolism and nutrition disorders) | 11 (13) | 9 (10) | 6 (10) | 3 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 62 (73) | 1 (1) | 16 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 27 (30) | 5 (7) | 11 (11)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 20 (24) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 11 (14) | 35 (44) | 2 (4) | 14 (18)
Insomnia (Psychiatric disorders) | 11 (11) | 39 (41) | 5 (5) | 11 (12)
Proteinuria (Renal and urinary disorders) | 13 (19) | 107 (184) | 11 (18) | 68 (120)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 46 (56) | 5 (6) | 14 (19)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 31 (35) | 3 (3) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 28 (29) | 2 (2) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 37 (45) | 2 (2) | 12 (12)
Alopecia (Skin and subcutaneous tissue disorders) | 22 (22) | 6 (6) | 7 (7) | 2 (2)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 76 (82) | 6 (7) | 33 (39) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 15 (16) | 71 (99) | 7 (8) | 24 (31)
Rash (Skin and subcutaneous tissue disorders) | 28 (28) | 46 (51) | 7 (7) | 21 (24)
Hypertension (Vascular disorders) | 38 (43) | 118 (191) | 12 (15) | 54 (90)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 17 (20) | 0 (0) | 9 (11)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 11 (14) | 1 (1) | 9 (12)
Malaise (General disorders) | 5 (5) | 13 (13) | 3 (3) | 6 (6)
Pain (General disorders) | 1 (1) | 9 (10) | 1 (1) | 9 (10)
Hepatic function abnormal (Hepatobiliary disorders) | 4 (4) | 8 (8) | 3 (3) | 8 (9)
Bilirubin conjugated increased (Investigations) | 4 (7) | 12 (28) | 6 (10) | 13 (29)
Blood bilirubin unconjugated increased (Investigations) | 1 (1) | 7 (19) | 2 (2) | 7 (19)
Blood lactate dehydrogenase increased (Investigations) | 7 (10) | 10 (14) | 9 (13) | 10 (13)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 10 (16) | 0 (0) | 11 (15)
Gamma-glutamyltransferase increased (Investigations) | 7 (7) | 11 (13) | 9 (9) | 16 (18)
Lymphocyte count decreased (Investigations) | 2 (4) | 15 (25) | 3 (5) | 9 (17)
Neutrophil count decreased (Investigations) | 5 (15) | 16 (46) | 5 (6) | 18 (56)
Protein urine present (Investigations) | 4 (4) | 3 (5) | 5 (5) | 5 (9)
Prothrombin time prolonged (Investigations) | 1 (1) | 6 (7) | 1 (1) | 7 (10)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 1 (1) | 8 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (10) | 3 (3) | 3 (3)
Cylindruria (Renal and urinary disorders) | 0 (0) | 7 (20) | 0 (0) | 8 (21)
Haematuria (Renal and urinary disorders) | 0 (0) | 13 (25) | 0 (0) | 8 (19)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 3 (3) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (6) | 10 (11) | 3 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT03434379/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT03434379/SAP_001.pdf